CLINICAL TRIAL: NCT07279818
Title: Effectiveness of Transcutaneous Acupoints Electrical Stimulation and Auricular Acupressure on Chemotherapy Induced Peripheral Neuropathy in Children With Leukemia: a Single Blind Randomized Controlled Study
Brief Title: Improving Chemotherapy Induced Peripheral Neuropathy in Children With Leukemia: A Study of Transcutaneous Acupoints Electrical Stimulation and Auricular Acupressure Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAES and AA to treat CIPN
Record Dates: First submitted 2025-11-22; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Keywords: Transcutaneous Acupoints Electrical Stimulation; Auricular Acupressure; chemotherapy induced peripheral neuropathy; Leukemia; children
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous Acupoints Electrical Stimulation (TAES) (Experimental): The intervention for TAES group will last 8 weeks, conducting 2 times per week, total covering 16 sessions. The intervention will be delivered a registered nurse with qualified TCM nurse certification. Four bilateral acupoints - Hegu, Shousanli , Zusanli, and Chongyang will be choosen. TAES will be deliveried by electronic acupunture treatment instrument with low frequency. Each session is 60 minutes.
  Interventions: Behavioral: Transcutaneous Acupoints Electrical Stimulation (TAES)
- Auricular Acupressure (AA) (Experimental): The AA subjects received auricular acupressure three times a day for two days every week for 8 weeks, total covering 16 sessions. Four acupoints including Shenmen (TF4), sympathetic (AH6a), fingers (SF1) and toes (AH2) will be choosen. A small piece of adhesive tape with vaccaria seed will be taped onto each selected auricular acupoint on a subject's ear.
  Interventions: Behavioral: Auricular Acupressure (AA)
- Self-Managed control group (Placebo Comparator): Subjects shall receive leaflet containing self-help materials for CIPN which they can conduct by themself (self-management) and continue to receive their usual care from the hospital.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Transcutaneous Acupoints Electrical Stimulation (TAES) — Transcutaneous Acupoints Electrical Stimulation (TAES) is a kind of physical therapy that use electric current through the electrodes placed on the surface of acupoints to produce clinical effects in the human body.
  Arms: Transcutaneous Acupoints Electrical Stimulation (TAES)
Behavioral: Auricular Acupressure (AA) — Auricular acupressure (AA) is a non-invasive therapy rooted in Traditional Chinese Medicine (TCM) that involves applying pressure to specific acupoints on the ear using Vaccaria seeds.
  Arms: Auricular Acupressure (AA)
Other: No intervention — No intervention
  Arms: Self-Managed control group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of Transcutaneous Acupoints Electrical Stimulation (TAES) and Auricular Acupressure (AA) on subject CIPN symptoms, sensory function, motor and physical function, psychological, physical symptoms and quality of life outcomes in Children with Leukemia.

The main questions it aims to answer are:

1. Does TAES and AA can improve CIPN symptoms, sensory function, motor and physical function, psychological, physical symptoms and quality of life outcomes in children with Leukemia compared with self-management control group?
2. Does TAES yield improvements in CIPN symptoms, sensory function, motor and physical function, psychological, physical symptoms and quality of life outcomes that are comparable to those achieved through AA in children with leukemia?

This proposed research is designed to conduct a three-arm RCT comparing TAES, AA to usual care in children with leukemia.

Subjects in TAES group will receive 8 weeks TAES on four acupoints. Subjects in AA group will receive 8 weeks on four acupoints. Subjects in self-management control group will receive usual care they will receive from the hospital. These three groups will be provided with a leaflet containing self-help materials for CIPN.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 17 years old
* diagnosed with leukemia
* received neurotoxic chemotherapy
* have developed score 9 or above CIPN symptoms according to Pediatric Chemotherapy-Induced Neuropathy (P-CIN)
* able to communicate and read Chinese

Exclusion Criteria:

* receiving multiple cancer treatment
* had a diagnosis of cancer in the central nervous system cancer, cancer relapse or secondary cancer
* having other neuromuscular disorders, for example, traumatic brain injury and cerebral palsy
* having other systematic diseases that cause toxicity in the peripheral nervous system, such as sickle cell disease (SCD), Guillain-Barre ́ Syndrome (GBS), anterior cutaneous nerve entrapment syndrome (ACNES), obstetric brachial plexus injury (OBPI), type I diabetes mellitus, postherpetic neuralgia (PHN), peroneal nerve injury, and reflex sympathetic dystrophy (RSD)
* acupoints areas with injuries, wounds or allodynia
* participated in any other CIPN non-pharmacological intervention programme
* having any impaired bone marrow suppression, liver or renal function
* contraindications to TEAS or auricular acupressure: such as having a pacemaker, skin infection, damage, or allergy to the electrodes
* suffering from mental illness or using antipsychotic drugs
* parents and children refused to give consent.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
CIPN severity - Pediatric Chemotherapy-Induced Neuropathy (P-CIN) | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  To evaluate the severity of CIPN. The Pediatric Chemotherapy-Induced Neuropathy scale contains 13 items, with eight items to rate CIPN symptoms in the hands and feet and five items to rate the difficulty of performing functional tasks. The total score ranges from 0 to 65 with higher scores indicating more severe CIPN.

SECONDARY OUTCOMES:
Sensory function outcomes | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Touch sensation were measured using monofilament examination with the best of both 2 trials on each side averaged.
Sensory function outcomes | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Vibration sensation were measured using a 128 Hz tuning fork, with the best of both 2 trials on each side averaged.
Motor and physical function | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Timed Up and Go test (TUG) will be used to evaluate the motor and physical function in children with leukemia.
Motor and physical function | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  30-second sitting-rising test will be used to evaluate the motor and physical function in children with leukemia.
Motor and physical function | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Handheld grip strength meter will be used to evaluate the motor and physical function in children with leukemia.
Psychological distress | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  National Comprehensive Cancer Network (NCCN) distress thermometer will be used to evaluate the psychological distress of children with leukemia. It included two parts: one is a single-item DT screening tool using an 11-point visual scale for respondents to rate their level of subjective distress from 0 (no distress) to 10 (extreme distress). A cut off value ≥4 was recommended to indicate a distressed patient; another is a 40-items problem list to identify potential sources of distress including practical, family, emotional, physical, and spiritual distress.
Physical symptoms | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  The therapy-related symptom checklist for children (TRSC-C) Chinese version will be used to assess the physical symptoms severity. The total TRSC-C score ranges between 0 to 120, with higher scores indicating greater severity of symptoms.
Quality of life outcome | Baseline, immediately after intervention (T1), 1 month after intervention (T2), and 3 month after intervention (T3)
  Pediatric Quality of Life Inventory version 3.0 cancer module (PedsQL 3.0 cancer module) will be used to evalute the quality of life for children with leukemia. The scale score was the average of the total item scores, with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No